CLINICAL TRIAL: NCT05100134
Title: Managed Access Programs for LDK378, Ceritinib
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLDK378A2401
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Anaplastic Lymphoma Kinase (ALK)- Positive Tumors; Non-small Cell Lung Cancer (NSCLC)
Keywords: MAP; Manage access program; ceritinib; ALK positive tumors; Non-small cell lung cancer (NSCLC); Anaplastic large cell lymphoma (ALCL); Inflammatory myofibroblastic tumour (IMT),; LDK378
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lymphoma, Large-Cell, Anaplastic; Granuloma, Plasma Cell | interventions — ceritinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: ceritinib — Patients receive ceritinib
  Other Names: LDK378

SUMMARY:
The purpose of this registration is to list Managed Access Programs (MAPs) related to LDK378, Ceritinib.

DETAILED DESCRIPTION:
CLDK378A2401 - No longer available - Managed Access Program (MAP) to provide access to Ceritinib, for ALK Positive Tumors.

CLDK378A2402 - No longer available - An open-label, multi-center, Expanded Treatment Protocol (ETP) of oral LDK378 in adult patients with non-small cell lung cancer (NSCLC) characterized by ALK positivity.

CLDK378A2003M - Available - Managed Access Program (MAP) Cohort Treatment Plan CLDK378A2003M to provide access to LDK378 (ceritinib), for ALK-Positive Tumor Pediatric Patients.

ELIGIBILITY:
Inclusion Criteria:

1. An independent request was received from a licensed physician.
2. The patient has a serious or life-threatening disease or condition and there is no comparable or satisfactory alternative therapy available for diagnosis, monitoring, or treatment.
3. The patient is not eligible or able to enroll in a clinical trial or continue participation in such trial.
4. There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
5. The patient must meet any other medical criteria established by the medical experts responsible for the product or by the health authority in the country of request (as applicable).
6. Provision of the product will not interfere with the initiation, conduct, or completion of a Novartis clinical trial or overall development program.
7. Managed Access provision is allowed per local laws/regulations.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult